CLINICAL TRIAL: NCT04911595
Title: Evaluation de l'Ischemie Musculaire au Cours de l'Artériopathie Oblitérante Des Membres Inférieurs
Brief Title: Evaluation of Muscle Ischemia in Arterial Claudication (Tsingtao)
Acronym: Tsingtao
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: CE-2018/109
Record Dates: First submitted 2020-08-25; First posted 2021-06-03 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-06

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: exercise oximetry — transcutaneous oxygen pressure is measured at the skin level on chest , buttocks and calves during a walking test 3.2 km*:h 10% slope. From the test result the decrease from rest of oxygen pressure (DROP) index is calculated to estimate muscle ischemia
Diagnostic Test: thallium scintigraphy — Muscle thallium fixation is measured immediately after a walking test 3.2 km*:h 10% slope and at 4 hours after the test. From the test result the difference of late and early radioactivity is calculated at the buttock and calf level and normalized to total body radioactivity to estimate muscle ischemia

SUMMARY:
The goal is to compare the results observed in patients that had both an exercise oximetry and a thallium scintigraphy for lower limb claudication

DETAILED DESCRIPTION:
On our routine pratice, patients suffering claudication (specifically atypical claudication or claudication of doubful vascular origin) have exercise oximetry to prove the vascular origin of pain. If still doubtful (inconsistency of pain and oximetry results) patients are referred for thallium scintigraphy. Our goal is to compare the results issued from these two test

ELIGIBILITY:
Inclusion Criteria:

* Claudication suspected of arterial origin

Exclusion Criteria:

* missing endopoint value

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for claudication of suspected arterial
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2010-06 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Correlation of thallium scintigraphy to oximetry results | 1 year
  The coefficient of correlation of DROP values to normalized late to early changes in radioactivity wil be calculated at the calf and buttock level

CONTACTS AND LOCATIONS:
Overall Officials: pierre abraham, MD; PhD, Principal Investigator — UH Angers
Locations (1):
- Centre hospitalier universitaire, Angers, France

IPD SHARING:
Plan to Share IPD: Undecided